CLINICAL TRIAL: NCT03188718
Title: Validation Study of the WatchPAT 200 in the Diagnosis of Obstructive Sleep Apnea in Children 4-12 Years of Age
Brief Title: WatchPAT Device Validation Study Compared to Polysomnography
Acronym: WPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Kaiser Permanente (Other); Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-0827
Record Dates: First submitted 2017-06-01; First posted 2017-06-15 (Actual); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Sleep Apnea Syndromes; Sleep Disorder; Sleep
Keywords: Polysomnogram; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Wake Disorders

STUDY DESIGN:
Masking Description: Blinded to the subject's diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- WatchPAT Intervention (Other): Wearing the WatchPAT device simultaneously while receiving a clinically indicated sleep study (polysomnogram).
  Interventions: Device: WatchPAT Intervention

INTERVENTIONS:
Device: WatchPAT Intervention — Wearing the device during their clinically indicated sleep study. This is a validation study to the gold-standard polysomnogram.

SUMMARY:
Validation study of a novel sleep Device compared to a traditional sleep study.

DETAILED DESCRIPTION:
This is an investigator-initiated validation study for the WatchPAT 200 device compared to the gold standard polysomnography procedure (sleep study). To evaluate the accuracy of the WatchPAT device compared to an in-laboratory Polysomnogram (PSG), measurements including obstructive apnea hypopnea index (OAHI), apnea hypopnea index (AHI), oxygen desaturation index (ODI) and other relevant sleep parameteres and indices will be compared. Ultimately, the diagnostic agreement of the WatchPAT device in detecting between normal sleep and mild sleep apnea architecture will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 5 through 12 years of age.
2. Referral to the Sleep Lab due to concerns for Obstructive Sleep Apnea (OSA) and presenting with symptoms such as:

   * snoring,
   * witnessed apneas,
   * daytime sleepiness, and
   * mouth breathing, etc.
3. Informed consent obtained.

Exclusion Criteria:

1. Medical conditions that can affect the tonometer reading such as:

   * peripheral vascular disease,
   * cyanotic heart disease,
   * systemic hypertension, and
   * sickle cell crisis.
2. Medical conditions that can potentially limit tolerance of the WatchPAT 200 device such as:

   * autism spectrum disorder,
   * Trisomy 21, and
   * neurodevelopmental disorders.
3. History of neuromuscular malformation
4. History of current supplemental oxygen use
5. History of current vasoactive, cardiac or seizure medication use
6. Inability or unwillingness to provide informed consent

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Sobremonte-King, MD, Principal Investigator — University of Colorado, Denver; Ann Halbower, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WatchPAT Intervention
Started | 45
Completed | 37
Not Completed | 8
Not completed — Participant noncompliance | 4
Not completed — Withdrawal by Subject | 1
Not completed — Device failure | 3

BASELINE CHARACTERISTICS:
Population: The 8 participants who did not complete the study are excluded from the baseline characteristics data.
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 19
  More than one race | 11
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Peripheral Arterial Tone Apnea-hypopnea Index (PAHI)
Description: Compare the results to the subjects clinical sleep study results. The PAHI measures presence of sleep apnea. Scores are counts of respiratory events per hour. A score of more than 2 indicates obstructive sleep apnea. Mild = 2-4.9, Moderate = 5-9.9, Severe = 10 or more.
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: events per hour
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
events per hour | 13.3 [3.1 to 63.4]

2. Secondary Outcome: Peripheral Arterial Tone Respiratory Disturbance Index (PRDI)
Description: Peripheral index from the device sensor as measured on the skin, similar to a pulse oximeter. Count of respiratory events that do not meet the criteria for apnea, but that cause a disturbance in sleep.
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: events per hour
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
events per hour | 18.3 [7.5 to 93]

3. Secondary Outcome: Oxygen Desaturation Index (ODI)
Description: Peripheral index from the device sensor similar to a pulse oximeter. Number of desaturations by 3 percent in 1 hour.
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: events per hour
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
events per hour | 4.9 [.3 to 43.3]

4. Secondary Outcome: Sleep Staging: Light and Deep
Description: Overall sleep architecture parameters as reported on the Sleep Study PSG final report. Includes hyponogram that outlines the percentage of total sleep time spent in each stage of sleep (N1, N2, N3-4, and REM).
Time Frame: Up to 10 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
minutes
  Light | 180 (48.5)
  Deep | 108 (35.3)

5. Secondary Outcome: Oxygen Saturation
Description: Amount of oxygen present in the subjects blood via pulse oximetry.
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: percentage of O2
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
percentage of O2 | 94 [90 to 95]

6. Secondary Outcome: Heart Rate
Description: Documentation of the Subjects heart rate.
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: beats per minute
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
beats per minute | 78 [52 to 104]

7. Secondary Outcome: Body Position
Description: Body position of sleeping subject to reflect upon overall sleep hygiene such as prone, supine, back, stomach, etc.
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
minutes
  Supine | 162 [0 to 489]
  Non-supine | 229 [0 to 434]

8. Secondary Outcome: Sleep Time (Total)
Description: The Total Sleep Duration time in minutes as recorded by the PSG.
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
minutes | 427 [155 to 515]

9. Secondary Outcome: Sleep Staging: REM
Description: as for outcome 4
Time Frame: Up to 10 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | WatchPAT Intervention
Number analyzed (Participants) | 37
minutes | 93.5 [27 to 276]

ADVERSE EVENTS:
Time Frame: Up to 10 hours
Arm/Group | WatchPAT Intervention
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03188718/Prot_SAP_000.pdf